CLINICAL TRIAL: NCT05540613
Title: Tai Chi Versus Conventional Exercise to Improve Cognitive Performance in Older Adults With Mild Cognitive Impairment (MCI): A Comparative Randomized Controlled Trial
Brief Title: Tai Chi Versus Conventional Exercise to Improve Cognitive Performance in Older Adults With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TC_MCI_RCT
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Education (Sham Comparator): A 26 weeks brain health and general health education program with two 1.5-hour sessions weekly.
  Interventions: Behavioral: Health Education
- Conventional Exercise (Active Comparator): A 26 weeks Conventional Exercise training with two 1.5-hour sessions weekly.
  Interventions: Behavioral: Conventional Exercise
- Tai Chi (Experimental): A 26 weeks Tai Chi training with two 1.5-hour sessions weekly.
  Interventions: Behavioral: Tai Chi

INTERVENTIONS:
Behavioral: Health Education — A 26 weeks brain health and general health education program with two 1.5-hour sessions weekly.
  Arms: Health Education
Behavioral: Conventional Exercise — A 26 weeks Conventional Exercise training with two 1.5-hour sessions weekly.
  Arms: Conventional Exercise
Behavioral: Tai Chi — A 26 weeks Tai Chi training with two 1.5-hour sessions weekly.
  Arms: Tai Chi

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of Tai Chi and conventional exercise on improving cognitive function in older adults with mild cognitive impairment (MCI). Participants will be randomized into three six-month programmes, namely Health Education group, Tai Chi group and Conventional Exercise group. Assessments will be conducted at baseline, after the 26-week interventions, and 26-week after the competition of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chinese older adults aged equal or larger than 50 years
* Ethnic Chinese
* MCI under criteria of Mayo Clinic, including the following

  i. people with subjective complaint about a decline in cognitive function. ii. total score in the Montreal Cognitive Assessment is equal or below the 7th percentile of the age- and education- corrected normative data of Hong Kong. iii. the decline in cognitive function does not impair daily functioning, as revealed by getting ≥2 marks in every item on the Chinese Lawton Instrumental Activities of Daily Living 4-point Scale).

Exclusion Criteria:

* medical history of major chronic diseases such as cancer, stroke, cerebro- and cardio-vascular diseases, and renal disease
* uncontrolled diabetes
* diagnosed with dementia or using anti-dementia medication
* diagnosed with psychiatric diseases or using psychiatric medication
* with diseases or on medications known to severely affect cognitive performance
* somatic condition (e.g., limb lost) that prevent participation in exercise
* impaired mobility by chronic diseases (e.g., neurological, musculoskeletal and autoimmune diseases)
* incapable to perform physical exercise
* regular exercise habit (>3 times 60-min Tai Chi or moderate-intensity conventional exercise weekly) in the past 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The score of the Montreal Cognitive Assessment (MoCA) | 26 weeks
  Change in the score of the Montreal Cognitive Assessment. The score ranged from 0 to 30. Higher score indicates a better cognitive function.
  Participants scoring equal or below the 7th percentile of the age- and education-corrected normative data will be considered as having MCI.
The score of the Montreal Cognitive Assessment (MoCA) | 52 weeks
  Change in the score of the Montreal Cognitive Assessment. The score ranged from 0 to 30. Higher score indicates a better cognitive function.
  Participants scoring equal or below the 7th percentile of the age- and education-corrected normative data will be considered as having MCI.

SECONDARY OUTCOMES:
Clinical Dementia Rating | 26 weeks and 52 weeks
  The Clinical Dementia Rating (CDR) is a numeric scale of 0-3 points based on clinician/ certified rater ratings of cognition and daily function in the domains of memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Rating from 0, 0.5, 1, 2 and 3 indicated subjects' cognitive function having healthy, very mild impairment, mild impairment, moderate impairment and severe impairment respectively.
Neurocognitive Test | 26 weeks and 52 weeks
  The NIH Toolbox Cognitive Function Battery (CFB) will be used to objectively evaluate the various cognitive domains. CFB assesses cognitive abilities in different cognitive domains, including memory, executive function and attention. CFB will be delivered on a tablet computer.
Subjective Cognitive Performance | 26 weeks and 52 weeks
  The Cognitive Self-Report Questionnaire (CSRQ) will be used to examine the subjective cognitive performance. The CSRQ is validated in Hong Kong and comprises 25 questions with an overall score ranging from 0-100. A higher score indicates worse self-perception on cognitive performance.
Subjective Memory complaints | 26 weeks and 52 weeks
  The memory inventory for the Chinese - a questionnaire exploring subjective memory complaints and the effects on daily activities - will be performed to examine the subjective memory complaints.
Subjective Sleep Quality | 26 weeks and 52 weeks
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quantity and the perceived restfulness and disturbance of sleep by gathering information on usual bed time, wake time, time to fall asleep, time of actual sleep, and quality of sleep. Each item is rated on a "0-3" Likert scale, with a higher score indicating poorer sleep quality.
The Hospital Anxiety and Depression Scale | 26 weeks and 52 weeks
  The Hospital Anxiety and Depression Scale assesses the severity of depression and anxiety. This 14-item questionnaire has subscales for both depression and anxiety and the overall score ranges from 0-21, with a higher score indicating more severe depressive/anxious symptoms.
The 12-Item Short Form Survey | 26 weeks and 52 weeks
  The 12-Item Short Form Survey measures health-related quality of life. It has 12 items assessing physical functioning, emotional and mental health, bodily pain, general health, vitality, and social functioning, with higher overall scores indicating a better quality of life.
Medication Use | 26 weeks and 52 weeks
  Subjects' use of medications, unrelated to dementia and psychiatric conditions (e.g., sleep, dyslipidemic and hypertensive pills) will be recorded along with detailed usage information. Data on medication dose and weekly frequency will be presented as the total number of lowest recommended dose in 7 days for the analysis.
Short Physical Performance Battery (SPPB) Test | 26 weeks and 52 weeks
  Physical function and balancing performance will be assessed using the Short Physical Performance Battery (SPPB). The SPPB involves repeated timed chair stands, timed standing balance (with feet in parallel in semi-tandem and tandem positions), and a 4-meter walk to measure the usual gait speed.
Habitual Physical Activity | 26 weeks and 52 weeks
  Actigraph/IPAQ method to monitor and record habitual physical activity. Actigraph activity monitor (wGT3X-BT or GT9X, Actigraph, USA), a 3-axis accelerometer, will be used to objectively determine the habitual daily physical movement/activities.

CONTACTS AND LOCATIONS:
Overall Officials: Parco Siu, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No